CLINICAL TRIAL: NCT03424993
Title: Vascular Effects of Dietary Salt in Humans With Salt-Resistant Blood Pressure: Dietary Counseling Study
Brief Title: Vascular Effects of Dietary Salt in Humans With Salt-Resistant Blood Pressure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, William Farquhar, Professor, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1083986
Record Dates: First submitted 2018-01-29; First posted 2018-02-07 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Healthy
Keywords: Endothelium, vascular; Cardiovascular Disease; Hemodynamics; Oxidative Stress; Dietary Sodium; Dietary Counseling
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary Sodium Restriction (Experimental): Daily habitual dietary sodium intake < 2000mg
  Interventions: Other: Dietary Sodium Restriction
- Control (Sham Comparator): Routine habitual dietary sodium intake >3400mg
  Interventions: Other: Control

INTERVENTIONS:
Other: Dietary Sodium Restriction — A registered dietician will counsel participants to reduce daily habitual dietary salt intake below 2000mg over 4 weeks
  Arms: Dietary Sodium Restriction
Other: Control — Participants will consume their routine habitual dietary sodium intake > 3400mg per day with regular pre determined check in phone calls from a registered dietician.
  Arms: Control

SUMMARY:
The purpose of this study is to determine the effects of dietary salt restriction on central hemodynamics and vascular function in men and women with salt resistant blood pressure.

DETAILED DESCRIPTION:
Cardiovascular disease remains a major Public Health problem and is the leading cause of death in the US. Dietary sodium restriction is considered an important lifestyle modification for individuals with hypertension; however, there is controversy about the effects of dietary salt given that many individuals do not have "salt sensitive" blood pressure. Deleterious effects of salt on the vasculature may explain the finding that chronic DSR reduces the cardiovascular event rate by 25%despite only minor reductions in BP. It is not known whether dietary sodium restriction improves central pulsatile hemodynamics, known to be related to the development of left ventricular hypertrophy and heart failure risk, and whether the hypothesized improvements in central hemodynamics are similar in men & women. The purpose of this study is to determine the effects of dietary sodium restriction through dietary counseling on central hemodynamics and vascular function in men and women with salt resistant blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Habitual dietary sodium intake > 3400mg per day

Exclusion Criteria:

* Abnormal resting ECG
* Current abnormal blood panel (assessed by comprehensive metabolic panel, lipid panel and complete blood count).
* Hypertension (currently taking anti-hypertensive medications or resting blood pressure >140/90 mmHg)
* Medical history of cardiovascular disease, malignant cancer, diabetes or kidney disease
* Obesity (Body Mass Index > 30)
* Current pregnancy
* Unable to provide consent

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-01-21 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Reflected Pulse Wave Amplitude | Change from baseline at 4 weeks
  Late systolic pulsatile load on the left ventricle represented by reflected pulse wave amplitude; assessed by echocardiography combined with applanation tonometry.

SECONDARY OUTCOMES:
Microvascular Function | Change from baseline at 4 weeks
  Cutaneous microvascular dilatory response to local heating assessed by laser Doppler flowmetry coupled with intradermal microdialysis
Conduit Artery Endothelial Dependent Dilation | Change from baseline at 4 weeks
  Brachial artery flow mediated dilation assessed by duplex ultrasound
Arterial Stiffness | Change from baseline at 4 weeks
  Carotid - Femoral pulse wave velocity assessed by applanation tonometry
Forward pulse wave amplitude | Change from baseline at 4 weeks
  Central hemodynamic assessment of the forward pulse wave amplitude assessed by echocardiography combined with applanation tonometry.

CONTACTS AND LOCATIONS:
Overall Officials: William B Farquhar, PhD, Principal Investigator — University of Delaware; David G Edwards, PhD, Principal Investigator — University of Delaware; Shannon Lennon, PhD, Principal Investigator — University of Delaware
Locations (1):
- Department of Kinesiology and Applied Physiology, University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Undecided